CLINICAL TRIAL: NCT00416390
Title: The Effect of Lycopene on DNA Damage in Human Prostate
Brief Title: Lycopene in Treating Patients With Prostate Cancer or Benign Prostatic Hyperplasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000492778; UIC-1999-0489
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2007-10

CONDITIONS: Nonmalignant Neoplasm; Prostate Cancer
Keywords: benign prostatic hyperplasia; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Neoplasms; Prostatic Neoplasms; Prostatic Hyperplasia | interventions — Lycopene; Biopsy

INTERVENTIONS:
Dietary Supplement: lycopene
Other: laboratory biomarker analysis
Procedure: biopsy

SUMMARY:
RATIONALE: Chemoprevention is the use of certain substances to keep cancer from forming, growing, or coming back. Eating a diet high in lycopene, a substance found in tomatoes and tomato products, may keep cancer from forming or growing. Collecting and storing samples of blood from patients with cancer to study in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This randomized clinical trial is studying how well lycopene works in treating patients with prostate cancer or benign prostatic hyperplasia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the ability of prostatic tissue to accumulate doses of lycopene in patients with prostate cancer or benign prostate hyperplasia.
* Determine whether the steady state level of DNA oxidation in blood and prostate tissue is responsive to lycopene dosing.
* Investigate the effect of lycopene dosing on the lipid peroxidation marker malondialdehyde in serum.
* Assess the importance of measuring multiple DNA oxidation products as biomarkers of oxidative stress and its chemoprevention.
* Determine the significance of DNA oxidation products in blood as an indicator of oxidative stress in the prostate.
* Measure prostate and blood uptake of the chemoprevention agent lycopene.

OUTLINE: This is a randomized, double-blind, placebo-controlled study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral lycopene once daily for 3 weeks.
* Arm II: Patients receive oral placebo once daily for 3 weeks. In both arms, patients undergo biopsy to confirm diagnosis of prostate cancer or benign prostatic hyperplasia after 3 weeks of study therapy.

Blood samples are collected at baseline and before surgery for biomarker/laboratory studies.

PROJECTED ACCRUAL: A total of 120 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following:

  * Prostate cancer
  * Benign prostate hyperplasia
* High blood levels of prostate-specific antigen
* Enlarged prostate

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Ability of prostatic tissue to accumulate doses of lycopene
Responsiveness of steady state level of DNA oxidation in blood and prostate tissue to lycopene dosing
Effect of lycopene on lipid peroxidation marker malondialdehyde in serum
Importance of measuring multiple DNA oxidation products as biomarkers of oxidative stress and its chemoprevention
Significance of DNA oxidation products in blood as an indicator of oxidative stress in the prostate
Prostate and blood uptake of the chemoprevention agent lycopene

CONTACTS AND LOCATIONS:
Overall Officials: Richard B. van Breemen, PhD, Principal Investigator — University of Illinois at Chicago

REFERENCES:
- [Derived] van Breemen RB, Sharifi R, Viana M, Pajkovic N, Zhu D, Yuan L, Yang Y, Bowen PE, Stacewicz-Sapuntzakis M. Antioxidant effects of lycopene in African American men with prostate cancer or benign prostate hyperplasia: a randomized, controlled trial. Cancer Prev Res (Phila). 2011 May;4(5):711-8. doi: 10.1158/1940-6207.CAPR-10-0288. Epub 2011 Mar 23. PMID 21430075